CLINICAL TRIAL: NCT03005184
Title: Mechanism(s) Underlying Cardiovascular Effects of ARB/NEP Inhibition - Aim 2
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study is being redesigned and submitted as a new study.
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, Hugh J. Morgan Professor of Medicine and Pharmacology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB#161306
Record Dates: First submitted 2016-12-22; First posted 2016-12-29 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Heart Failure NYHA Class I; Heart Failure NYHA Class II; Heart Failure NYHA Class III
MeSH Terms: interventions — Valsartan; BID protein, human; Enalapril; sacubitril and valsartan sodium hydrate drug combination; icatibant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (12):
- S/V+Pla, S/V+I, Enal+Pla, Enal+I (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- S/V+Pla, Enal+I, S/V+I, Enal+Pla (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- S/V+Pla, Enal+Pla, Enal+I, S/V+I (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- S/V+I, S/V+Pla, Enal+I, Enal+P (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- S/V+I, Enal+Pla, S/V+Pla, Enal+I (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- S/V+I, Enal+I, Enal+Pla, S/V+Pla (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- Enal+Pla, S/V+Pla, S/V+I, Enal+I (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- Enal+Pla, S/V+I, Enal+I, S/V+Pla (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- Enal+Pla, Enal+I, S/V+Pla, S/V+I (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- Enal+I, S/V+Pla, Enal+Pla, S/V+I (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- Enal+I, S/V+I, S/V+Pla, Enal+Pla (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo
- Enal+I, Enal+Pla, S/V+I, S/V+Pla (Experimental): Enal indicated Enalapril 10 mg bid for seven days, and S/V indicates Sacubitril-Valsartan 200 mg bid for seven days. Pla indicates intravenous placebo given on the seventh day of treatment, whereas I indicates intravenous icatibant given on the seventh day of treatment. Each treatment period is separated by a three-week washout during which patients receive Valsartan 80 mg bid.
  Interventions: Drug: Valsartan 80 mg bid; Drug: Enalapril 10 mg bid; Drug: Sacubitril-Valsartan 200 mg bid; Drug: Icatibant; Drug: Placebo

INTERVENTIONS:
Drug: Valsartan 80 mg bid — oral medication during run-in and washout period
Drug: Enalapril 10 mg bid — oral medication
Drug: Sacubitril-Valsartan 200 mg bid — oral medication
Drug: Icatibant — intravenous medication
Drug: Placebo — intravenous medication

SUMMARY:
This study tests the hypothesis that endogenous bradykinin contributes to effects of a combined angiotensin receptor blocker/neprilysin inhibitor (LCZ696 or Entresto)

DETAILED DESCRIPTION:
Patients with heart failure (HF) with reduced ejection fraction who qualify for the study will undergo a three-week run-in period in which any prior angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker they were taking will be discontinued and they will be given valsartan 80 mg bid in a single-blind fashion. After the run-in, subjects will undergo four study periods in random order. During two study periods they will receive enalapril 10 mg bid and during two they will receive sacubitril/valsartan (LCZ696) 200 mg bid for seven days. On the seventh day or each period, subjects will complete a study day in which they are randomized to receive either the bradykinin B2 receptor blocker icatibant or placebo intravenously. Each study period will be separated by a three-week washout during which subjects receive valsartan 80 mg bid.

ELIGIBILITY:
Inclusion Criteria:

1. Stable patients with a reduced EF

   1. EF less than or equal to 40% (confirmed by echocardiogram within the last six months), and
   2. history of symptoms of New York Heart Association class I, II or III HF
   3. stable clinical symptoms including no hospitalizations for the last six months
   4. treatment with a stable dose of an ACEi or ARB and with a beta blocker (unless contraindicated or not tolerated) for at least four weeks
   5. treatment with a stable dose of an MR antagonist for at least four weeks unless not possible due to renal function or serum potassium.
2. For female subjects, the following conditions must be met:

   1. postmenopausal status for at least one year, or
   2. status post-surgical sterilization

Exclusion Criteria:

1. History of hypersensitivity or allergy to any of the study drugs, drugs of similar chemical classes, ACEi, ARBs, or NEPi, as well as known or suspected contraindications to the study drugs
2. History of angioedema
3. History of pancreatitis or known pancreatic lesions
4. History of decompensated HF within the last six months (exacerbation of chronic HF manifested by signs and symptoms that required intravenous therapy or hospitalization)
5. History of heart transplant or on a transplant list or with left ventricular assistance device
6. Symptomatic hypotension and/or a SBP<100 mmHg at screening or <90 mmHg during the study
7. Serum potassium >5.2 mmol/L at screening or >5.4 mmol/L during the study
8. Acute coronary syndrome, cardiac, carotid, or other major cardiovascular surgery, percutaneous coronary intervention, or carotid angioplasty within six months prior to screening
9. Coronary or carotid artery disease likely to require surgical or percutaneous intervention within six months of screening
10. History of serious neurologic disease such as cerebral hemorrhage, stroke, seizure, or transient ischemic attack within six months
11. History of ventricular arrhythmia with syncopal episodes
12. Symptomatic bradycardia or second- or third-degree atrioventricular block without a pacemaker
13. Presence of hemodynamically significant mitral and/or aortic valve disease, except mitral regurgitation secondary to LV dilatation
14. Presence of other hemodynamically significant obstructive lesions of the left ventricular outflow tract, including aortic and subaortic stenosis
15. Type 1 diabetes
16. Poorly controlled type 2 diabetes mellitus (T2DM), defined as a HgbA1c >9%
17. Hematocrit <35%
18. Impaired renal function (eGFR of <30mL/min/1.73 m2) as determined by the four-variable Modification of Diet in Renal Disease (MDRD) equation, where serum creatinine (Scr) is expressed in mg/dL and age in years:

    eGFR (mL/min/1.73m2)=175 • Scr-1.154 • age-0.203 • (1.212 if Black) • (0.742 if female)
19. Use of hormone-replacement therapy
20. Breast feeding and pregnancy
21. History or presence of immunological or hematological disorders
22. History of malignancy other than non-melanoma skin cancer
23. Diagnosis of asthma requiring use of inhaled beta agonist more than once a week
24. Clinically significant gastrointestinal impairment that could interfere with drug absorption
25. Impaired hepatic function [aspartate amino transaminase (AST) and/or alanine amino transaminase (ALT) >3.0 x upper limit of normal range]
26. Any underlying or acute disease requiring regular medication which could possibly pose a threat to the subject or make implementation of the protocol or interpretation of the study results difficult, such as arthritis treated with non-steroidal anti-inflammatory drugs
27. Treatment with chronic systemic glucocorticoid therapy within the last year
28. Treatment with lithium salts
29. History of alcohol or drug abuse
30. Treatment with any investigational drug in the one month preceding the study
31. Mental conditions rendering the subject unable to understand the nature, scope, and possible consequences of the study
32. Inability to comply with the protocol, e.g., uncooperative attitude, inability to return for follow-up visits, and unlikelihood of completing the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-09 (Estimated); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
change in systolic blood pressure | 7-hour period after 7-day intervention
change in plasma cGMP | 7-hour period after 7-day intervention

SECONDARY OUTCOMES:
heart rate | 7-hour period after 7-day intervention
renal plasma flow | 7-hour period after 7-day intervention
glomerular filtration rate | 7-hour period after 7-day intervention
change in diastolic blood pressure | 7-hour period after 7-day intervention
fractional excretion of sodium | 7-hour period after 7-day intervention
urine albumin-to-creatinine ratio | 7-hour period after 7-day intervention
brain natriuretic peptide (BNP) to N-terminal pro-BNP ratio | 7-hour period after 7-day intervention
plasminogen activator inhibitor-1 | 7-hour period after 7-day intervention
tissue plasminogen activator | 7-hour period after 7-day intervention
aldosterone | 7-hour period after 7-day intervention
urine cGMP | 7-hour period after 7-day intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No